CLINICAL TRIAL: NCT02840877
Title: The Impact of Alcohol Consumption on Tuberculosis Treatment Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Medical Research Council, South Africa (Other); Boston University (Other); University of Cape Town (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Stellenbosch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-34970; 1R01AI119037-01A1 (NIH)
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Results first posted 2023-08-14 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Tuberculosis; Alcohol Consumption; Treatment Adverse Effect
Keywords: tuberculosis culture; alcohol use
MeSH Terms: conditions — Tuberculosis; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DOT Adherence Monitoring (Other): Daily adherence monitoring by study-employed directly observed therapy (DOT) worker on weekdays throughout the course of TB therapy
  Interventions: Behavioral: DOT Adherence Monitoring

INTERVENTIONS:
Behavioral: DOT Adherence Monitoring — Study participants will meet with a study-employed DOT worker daily during weekdays throughout the course of their TB treatment

SUMMARY:
After HIV/AIDS, tuberculosis (TB) remains the second leading cause of death due to an infectious disease globally. Retrospective studies from many countries, including the United States and South Africa, have consistently reported that in addition to having a higher burden of TB disease, patients with problem alcohol use have worse TB treatment outcomes. This prospective study will attempt to clarify both behavioral and biologic causal mechanisms underlying the deleterious effects of problem alcohol use on TB treatment response.

DETAILED DESCRIPTION:
A major knowledge gap is the degree to which poor treatment outcomes in alcohol-abusing patients are due to noncompliance alone. Problem alcohol use impacts on retention in care and adherence to daily TB treatment. Poor medication adherence and increased default from TB care have been documented for patients consuming alcohol regularly in several countries. Yet there has been no research to identify reasons (beyond adherence) for these poorer outcomes among patients with problem alcohol use. A key barrier to understanding the persistent biologic effect of alcohol on TB disease is inadequate data on adherence, including detailed data on daily adherence (or number of missed doses of medication). Research combining better approaches to alcohol ascertainment and adherence monitoring is needed to advance understanding of the pathways by which alcohol use and TB disease interact.

Aim 1: To (i) examine the associations between problem alcohol use and TB treatment outcomes, and (ii) demonstrate that these associations persist independent of adherence to TB treatment.

Aim 2: To evaluate the effect of problem alcohol use on the pharmacokinetics (PK)/pharmacodynamics (PD) of TB drugs.

Aim 3: We will use existing samples and data and continue to collect samples and data to (A) evaluate Mtb diversity in host, its dynamics overtime and in a specific set of drug resistance, drug tolerance, virulence and immune regulator genes, for evidence of directional and diversifying selection. We will (B) also evaluate how Mtb diversity and genes under selection associate with time-to culture conversion (three consecutive weeks of negative growth) and negative treatment outcomes, adherence, HIV, diabetes mellitus (DM), and substance use. We will (C) leverage MIC and sequence data from TRUST. We will combine these with a large public Mtb MIC and WGS dataset enriched for high-level antibiotic resistance generated by studies that include the NIAID funded Harvard TB Centers of Excellence for Translational Research (CETR). We will train an in silico MIC predictor and probe interactions between mutations and the Mtb lineage on a genome-wide scale. The current TRUST investigators, as well as Dr. Maha Farhat, Harvard Medical School will oversee this aim.

Aim 4: A) To compare rates of dysglycemia (both hyperglycemia and hypoglycemia) in people living with HIV (PLWH) and HIV-uninfected persons receiving TB treatment in order to assess changes in blood glucose levels from study enrollment by HIV status and how alcohol use mediates the relationship; and B) to assess the role stress, inflammation and alcohol consumption play in relation to blood sugar levels in PLWH and HIV-uninfected individuals and to assess epigenetic modifications at DNA sites known to be involved in TB risk and neutrophil, monocyte, T and B cell function.

Culture-positive, pulmonary TB patients will be recruited in Worcester, South Africa, and followed over an 18-month period. Patients will complete an interviewer-administered questionnaire on their alcohol use and other health-related behaviors, and their recent alcohol use will be confirmed using a biomarker (phosphatidylethanol). Chest radiographs, sputum smears and culture, and blood samples will be collected to compare the biology of treatment response in patients with and without problem alcohol use. During the 6-month treatment period, smart mobile-phone technology will be used to document daily drug adherence by trained community workers. Serial measures of alcohol intake and serial sputa isolates will be collected to assess treatment response and TB drug side effects will be recorded. In addition, intensive PK/PD studies of isoniazid, rifampin, ethambutol, and pyrazinamide will be performed in 200 HIV-seronegative patients. The full cohort will be followed for 12 months post-treatment to examine long-term TB outcomes, including relapse and death.

ELIGIBILITY:
Inclusion Criteria:

1. at least 15 years old
2. initiating TB treatment in South Africa
3. expect to remain in the local area for the next 2 years
4. agree to comply with all study requirements, including provision of contact information and attendance at all study appointments
5. provide written, informed consent to participate in the study if ≥18 years of age or written assent and parental consent if <18 years.

Exclusion Criteria:

1. they have multidrug-resistant (MDR) TB (RIF resistance will be known at screening from Xpert MTB/RIF)
2. they have a contra-indication to start on standard 4-drug therapy
3. they are pregnant at study enrollment
4. they are HIV seropositive for aim 2 only

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2023-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Jacobson, MD MPH, Principal Investigator — Boston Medical Center, Department of Medicine
Locations (1):
- Worcester Community Day Centre, Worcester, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Overbeck V, Malatesta S, Carney T, Myers B, Parry CDH, Horsburgh CR, Theron D, White LF, Warren RM, Jacobson KR, Bouton TC. Understanding the impact of pandemics on long-term medication adherence: directly observed therapy in a tuberculosis treatment cohort pre- and post-COVID-19 lockdowns. BMC Infect Dis. 2024 Oct 14;24(1):1154. doi: 10.1186/s12879-024-09994-7. PMID 39396938
- [Derived] Ragan EJ, Gill CJ, Banos M, Bouton TC, Rooney J, Horsburgh CR, Warren RM, Myers B, Jacobson KR. Directly Observed Therapy to Measure Adherence to Tuberculosis Medication in Observational Research: Protocol for a Prospective Cohort Study. JMIR Res Protoc. 2021 Jun 16;10(6):e24510. doi: 10.2196/24510. PMID 34132642
- [Derived] Myers B, Bouton TC, Ragan EJ, White LF, McIlleron H, Theron D, Parry CDH, Horsburgh CR, Warren RM, Jacobson KR. Impact of alcohol consumption on tuberculosis treatment outcomes: a prospective longitudinal cohort study protocol. BMC Infect Dis. 2018 Sep 29;18(1):488. doi: 10.1186/s12879-018-3396-y. PMID 30268101

RESULTS

PARTICIPANT FLOW:
Groups:
- TRUST Cohort: TRUST Study Cohort
Period: Baseline to 12 Weeks
Arm/Group | TRUST Cohort
Started | 303
Completed | 282
Not Completed | 21
Not completed — Withdrawal by Subject | 11
Not completed — Moved/Transferred out | 5
Not completed — Lost to Follow-up | 2
Not completed — Death | 1
Not completed — Changed treatment regimen, no longer on first line drugs. | 1
Not completed — Treatment extended due to bacterial meningitis. | 1
Period: 12 Weeks to 6 Months
Arm/Group | TRUST Cohort
Started | 282
Completed | 271
Not Completed | 11
Not completed — Withdrawal by Subject | 4
Not completed — Treatment failure | 1
Not completed — Moved/transferred out | 1
Not completed — Lost to Follow-up | 4
Not completed — Death | 1
Period: 6 Months to 18 Months
Arm/Group | TRUST Cohort
Started | 271
Completed | 205
Not Completed | 66
Not completed — Withdrawal by Subject | 1
Not completed — Treatment failure | 7
Not completed — Relapse/recurrence of TB | 8
Not completed — Moved/transferred out | 6
Not completed — Lost to Follow-up | 24
Not completed — Death | 4
Not completed — Diagnosed with multi-drug resistant tuberculosis. | 1
Not completed — Treatment stopped due to liver injury. | 1
Not completed — Still in study. | 14

BASELINE CHARACTERISTICS:
Arm/Group | TRUST Cohort
Number analyzed (Participants) | 303
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [27 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121
  Male | 182
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Coloured/Mixed Ancestry | 284
  Black African | 16
  Indian/Asian | 1
  Other | 2
Region of Enrollment [Number; unit: participants]
  South Africa | 303

OUTCOME MEASURES:

1. Primary Outcome: Time to Culture Conversion
Description: Time to sterilization/culture conversion during the first twelve weeks of treatment in patients with problem alcohol use compared to those without
Time Frame: 12 weeks
Population: Individuals newly diagnosed with tuberculosis and initiating treatment were classified at baseline into either Low Alcohol Use (n=102), Moderate Alcohol Use (n=133), and High Alcohol Use (n=65). 3 participants were missing data on alcohol use as their baseline PEth tests were water damaged. Therefore the overall number of participants analyzed was 300 and the respective number of participants for each of the 3 levels of alcohol use are provided as just described.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | TRUST Cohort
Number analyzed (Participants) | 300
weeks
  Low Alcohol Use: number analyzed (Participants) | 102
  Low Alcohol Use | 5.6 (2.5)
  Moderate Alcohol Use: number analyzed (Participants) | 133
  Moderate Alcohol Use | 5.4 (2.5)
  High Alcohol Use: number analyzed (Participants) | 65
  High Alcohol Use | 5.5 (2.6)

2. Primary Outcome: Cmax
Description: Peak concentrations (Cmax) of isoniazid, rifampin, pyrazinamide, and ethambutol in patients with problem alcohol use compared to those without
Time Frame: 4 weeks
Population: Cmax outcome measure data was collected for 104 study participants who were enrolled into Aim 2 for pharmacokinetic/pharmacodynamic analysis. This measure was collected for 4 first-line TB medications: rifampicin, isoniazid, pyrazinamide, and ethambutol.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | TRUST Cohort
Number analyzed (Participants) | 104
mg/L
  Rifampicin | 5.29 [3.53 to 6.88]
  Isoniazid | 1.63 [1.25 to 2.23]
  Pyrazinamide | 28.5 [26.2 to 32.8]
  Ethambutol | 1.98 [1.75 to 2.20]

3. Primary Outcome: Area Under Curve (AUC)
Description: Individual patient steady state 24-hour area under curve (AUC) of isoniazid, rifampin, pyrazinamide, and ethambutol
Time Frame: 4 weeks
Population: AUC outcome measure data was collected for 104 study participants who were enrolled into Aim 2 for pharmacokinetic/pharmacodynamic analysis. This measure was collected for 4 first-line TB medications: rifampin, isoniazid, pyrazinamide, and ethambutol.
Measure: Median (Inter-Quartile Range); unit: mg x h/L
Arm/Group | TRUST Cohort
Number analyzed (Participants) | 104
mg x h/L
  Rifampin | 22.2 [15.5 to 31.2]
  Isoniazid | 6.32 [4.53 to 13.1]
  Pyrazinamide | 259 [236 to 292]
  Ethambutol | 13.2 [11.7 to 15.1]

4. Secondary Outcome: Poor Treatment Outcome
Description: Number and percent of participants that had favorable (defined as cured, treatment completed) and unfavorable (defined as treatmentfailure, death, relapse) TB outcomes. The 'other' category is defined as the treatment defaulted, was extended, participant moved or was transferred).
Time Frame: 18 months
Population: 3 individuals were excluded from overall numbers (total N=303) because they didn't have baseline Peth collected, so there did not have alcohol use data.
Measure: Count of Participants; unit: Participants
Arm/Group | TRUST Cohort
Number analyzed (Participants) | 300
Participants
  Favorable | 246
  Unfavorable | 24
  Other | 19
  Missing | 11

5. Secondary Outcome: Side Effects to TB Drugs
Description: Nember and percentage of patients who develop side effects to the TB drugs in patients with problem alcohol use compared to those without
Time Frame: 6 months
Population: 3 individuals were excluded from overall numbers (total N=303) because they didn't have baseline Peth collected, so they did not have alcohol use data
Measure: Count of Participants; unit: Participants
Arm/Group | TRUST Cohort
Number analyzed (Participants) | 300
Participants
  Side effects | 154
  No side effects | 146

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | TRUST Cohort
All-Cause Mortality (participants affected / at risk) | 8/303
Serious Adverse Events (participants affected / at risk) | 10/303
Other Adverse Events (participants affected / at risk) | 0/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRUST Cohort (N=303)
Participant death (General disorders) | 8 (8) — These deaths were unexpected and all were investigated and deemed unrelated to study participation. Total count may increase as 49 participants are still enrolled in the study.
Participant coughing up blood during transport (General disorders) | 1 (1) — Participant was referred to care and hospitalized. The incident was not related to study procedures. Total count may increase as 49 participants are still enrolled in the study.
Ineligible participant enrolled (Investigations) | 1 (1) — The participant was found to have extra-pulmonary TB during the enrollment visit, making them ineligible for the study. They were withdrawn and their samples were destroyed. Total count may increase as 49 participants are still enrolled in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT02840877/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT02840877/ICF_001.pdf